CLINICAL TRIAL: NCT00698607
Title: Comparison of the Efficacy of Everolimus-Eluting Versus Sirolimus-Eluting Stent for Coronary Lesions
Brief Title: Efficacy of Xience/Promus Versus Cypher in rEducing Late Loss After stENTing
Acronym: EXCELLENT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Abbott (Industry); Boston Scientific Corporation (Industry)
Responsible Party: Hyo-Soo, Kim, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXCELLENT
Record Dates: First submitted 2008-06-15; First posted 2008-06-17 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Coronary Artery Disease
Keywords: Everolimus; Sirolimus; drug eluting stent; Clopidogrel
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- E6 (Experimental): Everolimus-eluting stent 6-month clopidogrel therapy
  Interventions: Device: Everolimus-eluting stent (Xience or Promus); Drug: 6-month clopidogrel therapy
- S6 (Active Comparator): Sirolimus-eluting stent 6-month clopidogrel therapy
  Interventions: Device: Sirolimus-eluting stent (Cypher); Drug: 6-month clopidogrel therapy
- E12 (Experimental): Everolimus-eluting stent 12-month clopidogrel therapy
  Interventions: Device: Everolimus-eluting stent (Xience or Promus); Drug: 12-month clopidogrel therapy
- S12 (Active Comparator): Sirolimus-eluting stent 12-month clopidogrel therapy
  Interventions: Device: Sirolimus-eluting stent (Cypher); Drug: 12-month clopidogrel therapy

INTERVENTIONS:
Device: Everolimus-eluting stent (Xience or Promus) — Use everolimus-eluting stent in the treatment of coronary stenosis
  Other Names: Xience; Promus
  Arms: E12; E6
Device: Sirolimus-eluting stent (Cypher) — Use sirolimus-eluting stent in the treatment of coronary stenosis
  Other Names: Cypher
  Arms: S12; S6
Drug: 6-month clopidogrel therapy — Use clopidogrel for 6 months
  Other Names: Plavix
  Arms: E6; S6
Drug: 12-month clopidogrel therapy — Use clopidogrel for 12 months
  Other Names: Plavix
  Arms: E12; S12

SUMMARY:
Objectives

1. To evaluate the safety and long-term effectiveness of coronary stenting with the Everolimus-eluting coronary stent system(EECSS) (XIENCETM V, Abbott Vascular, Santa Clara, CA, PromusTM, Boston Scientific, Natick, MA), compared with the sirolimus-eluting coronary stent system(SECSS) (CypherTM, Cordis Johnson & Johnson, Warren, NJ) in the treatment of coronary stenosis.
2. To evaluate the safety and efficacy of 6-month clopidogrel therapy compared with 12-month clopidogrel therapy.

Study Design: Prospective, open label, two-arm, randomized multi-center trial to test the non-inferiority of EECSS compared with the SECSS, and to test the non-inferiority of 6 months duration compared with 12 months duration of clopidogrel therapy. Patients will be randomized in a two by two factorial manner according to the type of drug eluting stent (EECSS vs. SECSS) and the duration of dual anti-platelet therapy (6 months vs. 12 months). Randomization will also be stratified per hospital for the presence of DM and the presence of long lesions (lesion length ≥ 28mm)

Patient Enrollment: 1,372 patients enrolled at 17 centers in Korea.

Patient Follow-Up: Clinical follow-up will occur at 1, 3, and 9 months, and at 1, 2, 3, 4, and 5 years. Investigator or designee may conduct follow-up as telephone contacts or office visits.

Primary Endpoint

* In-segment late luminal loss (LL) at 9 months for comparison of stenting with EECSS vs. SECSS.
* Target vessel failure (TVF) (cardiac death, myocardial infarction, ischemia driven target vessel revascularization) at 12 months for comparison of 6 months vs. 12 months of clopidogrel therapy

Secondary Endpoint

* All Death
* Cardiac death
* Myocardial infarction
* Target vessel revascularization (TVR) (all and ischemia-driven)
* Target lesion revascularization (TLR) (all and ischemia-driven)
* Stent thrombosis
* Acute success (device, lesion, and procedure)
* Bleeding
* Cerebrovascular accident
* In-stent LL at 9 months
* Angiographic pattern of restenosis at 9-month angiographic follow-up
* In-stent and in-segment % diameter stenosis (%DS) at 9 months
* In-stent % volume obstruction (%VO) at 9 months
* Incomplete stent apposition post index procedure
* Persisting incomplete stent apposition, late-acquired incomplete stent apposition, aneurysm, thrombosis, and persisting dissection at 9 months

ELIGIBILITY:
General Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving the XIENCE V EECS and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
3. Subject must have significant coronary artery stenosis (>50% by visual estimate)
4. Subject must have evidence of myocardial ischemia (e.g., stable, unstable angina, recent infarction, silent ischemia, positive functional study or a reversible changes in the electrocardiogram (ECG) consistent with ischemia. In subjects with coronary artery stenosis > 75%, evidence of myocardial ischemia does not have to be documented.
5. Subjects must be an acceptable candidate for Coronary Artery Bypass Graft (CABG) surgery.

Angiographically Inclusion Criteria

1. Target lesion(s) must be located in a native coronary artery with visually estimated diameter of ≥ 2.25 mm and ≤ 4.25 mm.
2. Target lesion(s) must be amenable for percutaneous coronary intervention

General Exclusion Criteria:

1. The patient has a known hypersensitivity or contraindication to any of the following medications (heparin, aspirin, clopidogrel, sirolimus, everolimus, Contrast media
2. Systemic (intravenous) Sirolimus, everolimus use within 12 months.
3. Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
4. History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions.
5. Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months.
6. Current known current platelet count <100,000 cells/mm3 or Hgb <10 g/dL.
7. An elective surgical procedure is planned that would necessitate interruption of clopidogrel during the first 12 months post enrollment.
8. Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
9. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
10. Patients who have received any stent implantation in the target vessel prior to enrollment.
11. Patients with LVEF<25% or those with cardiogenic shock
12. Patients with myocardial infarction within 72 hours
13. Creatinine level ≥ 3.0mg/dL or dependence on dialysis.
14. Severe hepatic dysfunction (AST and ALT: 3 times upper normal reference values).

Angiographic Exclusion Criteria

1. Patients with significant left main coronary artery stenosis
2. Patients who's target lesion has in-stent restenosis at the stented segment of drug-eluting stents or bare metal stents
3. Target lesions with chronic total occlusion
4. True bifurcation lesions requiring two stents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1466 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
In-segment late luminal loss (LL) at 9 months for comparison of stenting with EECSS vs. SECSS. | 9 months
Target vessel failure (TVF) (cardiac death, myocardial infarction, ischemia driven target vessel revascularization) at 12 months for comparison of 6 months vs. 12 months of clopidogrel therapy | 12 months

SECONDARY OUTCOMES:
All death | 5 years
Cardiac death | 5 Years
Myocardial infarction | 5 years
Target vessel revascularization (TVR) (all and ischemia-driven) | 5 years
Target lesion revascularization (TLR) (all and ischemia-driven) | 5 years
Stent thrombosis | 5 years
Acute success (device, lesion, and procedure) | Index procedure
Bleeding | 5 years
Cerebrovascular accident | 5 years
In-stent LL at 9 months | 9 months
Angiographic pattern of restenosis at 9-month angiographic follow-up | 9 months
In-stent and in-segment % diameter stenosis (%DS) at 9 months | 9 months
In-stent % volume obstruction (%VO) at 9 months | 9 months
Incomplete stent apposition post index procedure | Index procedure
Persisting incomplete stent apposition, late-acquired incomplete stent apposition, aneurysm, thrombosis, and persisting dissection at 9 months | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, MD, PhD, Study Chair — Seoul National University Hospital; Yangsoo Jang, MD, PhD, Study Chair — Yonsei University; Jung-Han Yoon, MD, PhD, Study Chair — Yonsei Univercity Wonju hospital; Ahn Tae-Hoon, MD, PhD, Study Chair — Gachon Kil Medical Center; Hyun-Cheol Kwon, MD, PhD, Study Chair — Samsung Medical Center; In-Ho Chae, MD, PhD, Study Chair — Seoul National University Bundang Hospital; Young-Jin Choi, MD, PhD, Principal Investigator — Hallym University Medical Center; Kyoo-Rok Han, MD, PhD, Principal Investigator — Kandong Sacred heart Hospital; Si-Hoon Park, MD, PhD, Principal Investigator — Ewha Women's University Hospital; Myeong-Ho Chung, MD, PhD, Principal Investigator — Chonnam National University Hospital; Hyuk-Moon Kwon, MD, PhD, Principal Investigator — Yonsei University; Dong-Woon Chun, MD, PhD, Principal Investigator — National Health Insurance Service Ilsan Hospital; Byung-Ok Kim, MD, PhD, Principal Investigator — Inje University Sanggye Hospital; Do-Sun Lim, MD, PhD, Principal Investigator — Korea University Anam Hospital; Taek-Jong Hong, MD, PhD, Principal Investigator — Pusan National University Hospital; Woo-Young Chung, MD, PhD, Principal Investigator — Borame Hospital; Jae-Hun Chung, MD, PhD, Principal Investigator — Hallym University Kangnam Sacred Heart Hospital
Locations (1):
- Seoul National University Hospital, Seoul, 28 Yongon Dong, Jongro Gu, South Korea

REFERENCES:
- [Derived] Jang JY, Jung HW, Lee BK, Shin DH, Kim JS, Hong SJ, Ahn CM, Kim BK, Ko YG, Choi D, Hong MK, Park KW, Gwon HC, Kim HS, Kwon HM, Jang Y. Impact of PRECISE-DAPT and DAPT Scores on Dual Antiplatelet Therapy Duration After 2nd Generation Drug-Eluting Stent Implantation. Cardiovasc Drugs Ther. 2021 Apr;35(2):343-352. doi: 10.1007/s10557-020-07008-7. PMID 32588238
- [Derived] Kang J, Han JK, Kang DY, Zheng C, Yang HM, Park KW, Kang HJ, Koo BK, Kim HS. SYNTAX Score and SYNTAX Score II Can Predict the Clinical Outcomes of Patients with Left Main and/or 3-Vessel Disease Undergoing Percutaneous Coronary Intervention in the Contemporary Cobalt-Chromium Everolimus-Eluting Stent Era. Korean Circ J. 2020 Jan;50(1):22-34. doi: 10.4070/kcj.2019.0097. Epub 2019 Sep 30. PMID 31642213
- [Derived] Jang JY, Shin DH, Kim JS, Hong SJ, Ahn CM, Kim BK, Ko YG, Choi D, Hong MK, Park KW, Gwon HC, Kim HS, Jang Y. Optimal duration of DAPT after second-generation drug-eluting stent in acute coronary syndrome. PLoS One. 2018 Nov 26;13(11):e0207386. doi: 10.1371/journal.pone.0207386. eCollection 2018. PMID 30475845
- [Derived] Park KW, Rhee TM, Kang HJ, Koo BK, Gwon HC, Yoon JH, Lim DS, Chae IH, Han KR, Ahn T, Jeong MH, Jeon DW, Jang YS, Kim HS. Randomized Prospective Comparison of Everolimus-Eluting vs. Sirolimus-Eluting Stents in Patients Undergoing Percutaneous Coronary Intervention - 3-Year Clinical Outcomes of the EXCELLENT Randomized Trial. Circ J. 2018 May 25;82(6):1566-1574. doi: 10.1253/circj.CJ-17-0677. Epub 2017 Sep 30. PMID 28966335
- [Derived] Ko YG, Shin DH, Kim JS, Kim BK, Choi D, Hong MK, Gwon HC, Ahn T, Chae IH, Yoon JH, Kim HS, Jang Y; EXCELLENT investigators. Comparison of neointimal hyperplasia and peri-stent vascular remodeling after implantation of everolimus-eluting versus sirolimus-eluting stents: intravascular ultrasound results from the EXCELLENT study. Int J Cardiovasc Imaging. 2013 Aug;29(6):1229-36. doi: 10.1007/s10554-013-0199-5. Epub 2013 Mar 3. PMID 23456359
- [Derived] Gwon HC, Hahn JY, Park KW, Song YB, Chae IH, Lim DS, Han KR, Choi JH, Choi SH, Kang HJ, Koo BK, Ahn T, Yoon JH, Jeong MH, Hong TJ, Chung WY, Choi YJ, Hur SH, Kwon HM, Jeon DW, Kim BO, Park SH, Lee NH, Jeon HK, Jang Y, Kim HS. Six-month versus 12-month dual antiplatelet therapy after implantation of drug-eluting stents: the Efficacy of Xience/Promus Versus Cypher to Reduce Late Loss After Stenting (EXCELLENT) randomized, multicenter study. Circulation. 2012 Jan 24;125(3):505-13. doi: 10.1161/CIRCULATIONAHA.111.059022. Epub 2011 Dec 16. PMID 22179532
- [Derived] Park KW, Chae IH, Lim DS, Han KR, Yang HM, Lee HY, Kang HJ, Koo BK, Ahn T, Yoon JH, Jeong MH, Hong TJ, Chung WY, Jo SH, Choi YJ, Hur SH, Kwon HM, Jeon DW, Kim BO, Park SH, Lee NH, Jeon HK, Gwon HC, Jang YS, Kim HS. Everolimus-eluting versus sirolimus-eluting stents in patients undergoing percutaneous coronary intervention: the EXCELLENT (Efficacy of Xience/Promus Versus Cypher to Reduce Late Loss After Stenting) randomized trial. J Am Coll Cardiol. 2011 Oct 25;58(18):1844-54. doi: 10.1016/j.jacc.2011.07.031. PMID 22018294
- [Derived] Park KW, Yoon JH, Kim JS, Hahn JY, Cho YS, Chae IH, Gwon HC, Ahn T, Oh BH, Park JE, Shim WH, Shin EK, Jang YS, Kim HS. Efficacy of Xience/promus versus Cypher in rEducing Late Loss after stENTing (EXCELLENT) trial: study design and rationale of a Korean multicenter prospective randomized trial. Am Heart J. 2009 May;157(5):811-817.e1. doi: 10.1016/j.ahj.2009.02.008. PMID 19376305